CLINICAL TRIAL: NCT03480269
Title: Very Rapid and Rapid Virological Response as Predictors of Response to Sofosbuvir / Daclatasvir Treatment of HCV Related Liver Disease
Brief Title: Very Rapid and Rapid Virological Response as Predictors of Response of HCV Tretment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Mahrous Sayed, Doctor, Assiut University
Other Study IDs: HCV tretment
Record Dates: First submitted 2018-03-02; First posted 2018-03-29 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-03

CONDITIONS: Predictors of Response to HCV Tretment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assessment of very rapid virological response and rapid virological response as predictors of response to sofosbuvir and daclatasvir in treatment of cirrhotic and non-cirrhotic patients with HCV, eligible to treatment.

DETAILED DESCRIPTION:
Chronic hepatitis C infection (CHC) is a global health problem, with an estimated 120 to 130 million chronic hepatitis C virus (HCV) carriers worldwide Therefore, early recognition and effective management of the disease can modify its natural history

. There is a growing body of evidence that suggests that treatment will help reduce liver inflammation, may reverse liver damage (scarring),slow down disease progression and improve symptoms and quality of life. All of these factors are important reasons to seek HCV medical treatment Identifying host-viral factors that predict the likelihood of SVR prior to initiating therapy would be a very useful clinical tool that could help reduce costs and avoid unnecessary exposure to therapy with significant side effects Little is known about predictors of failure to achieve SVR with DAAs. Although numerous clinical parameters predicted poor response to pegylated IFN treatment , none of them have been shown to be associated with virological relapse after DAA based therapy

Treatment response terms:

The ultra rapid virological response (uRVR) is a new endpoint that we defined as an undetectable serum HCV RNA at the end of 1st week of therapy.

The very rapid virologic response( vRVR )defined as undetectable serum HCV RNA level at week 2.

The rapid virological response (RVR) defined as undetectable serum HCV RNA after 4 weeks of treatment sustained virological response (SVR), which is defined by the undetectable serum HCV RNA 12-24 weeks after the end of treatment Relapser was defined as undetectable viral load at the end of DAA treatment but subsequent detectable viral load at 12 weeks after treatment end.

ELIGIBILITY:
Inclusion Criteria:

* Anti HCV positive patients either chronic HCV or liver cirrhosis.
* Detectable HCV RNA by quantitative PCR prior to treatment.
* Naïve patients (not received any HCV treatment regimen before)

Exclusion Criteria:

* Patients with hepatocellular carcinoma( HCC)
* Patients with combined HBV and HCV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with HCV related liver disease ( either cirrhotic or non cirrhotic) eligible to tretment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Rapid virological response (undetected HCV RNA after 4 weeks from the begin of antiviral treatment) | April 2018 to April 2019
  To assess rapid virological response as a predictor of response to sofosbuvir and daclatasvir in treatment of cirrhotic and non-cirrhotic patients with HCV. It measure the relation between rapid virological response and achievment of sustained virological response (Undetected HCV RNA 12-24 weeks after the end of treatment )

REFERENCES:
- [Background] Patel K, Lucas JE, Thompson JW, Dubois LG, Tillmann HL, Thompson AJ, Uzarski D, Califf RM, Moseley MA, Ginsburg GS, McHutchison JG, McCarthy JJ; MURDOCK Horizon 1 Study Team. High predictive accuracy of an unbiased proteomic profile for sustained virologic response in chronic hepatitis C patients. Hepatology. 2011 Jun;53(6):1809-18. doi: 10.1002/hep.24284. Epub 2011 May 14. PMID 21381069
- [Background] Cavalcante LN, Lyra AC. Predictive factors associated with hepatitis C antiviral therapy response. World J Hepatol. 2015 Jun 28;7(12):1617-31. doi: 10.4254/wjh.v7.i12.1617. PMID 26140082
- [Background] Childs K, Merritt E, Considine A, Sanchez-Fueyo A, Agarwal K, Martinez-Llordella M, Carey I. Immunological Predictors of Nonresponse to Directly Acting Antiviral Therapy in Patients With Chronic Hepatitis C and Decompensated Cirrhosis. Open Forum Infect Dis. 2017 Apr 3;4(2):ofx067. doi: 10.1093/ofid/ofx067. eCollection 2017 Spring. PMID 28584852
- [Background] Yakoot M, Abdo AM, Yousry A, Helmy S. Very rapid virologic response and early HCV response kinetics, as quick measures to compare efficacy and guide a personalized response-guided therapy. Drug Des Devel Ther. 2016 Aug 25;10:2659-67. doi: 10.2147/DDDT.S111496. eCollection 2016. PMID 27601883
- [Background] Yek C, de la Flor C, Marshall J, Zoellner C, Thompson G, Quirk L, Mayorga C, Turner BJ, Singal AG, Jain MK. Effectiveness of direct-acting antiviral therapy for hepatitis C in difficult-to-treat patients in a safety-net health system: a retrospective cohort study. BMC Med. 2017 Nov 20;15(1):204. doi: 10.1186/s12916-017-0969-3. PMID 29151365